CLINICAL TRIAL: NCT06626594
Title: Reliability and Validity of the Chinese Version of the Neonatal Sleep-Wake Assessment Tool
Status: Withdrawn | Type: Observational
Why Stopped: This study, part of the NCT06573203 study, used the same ethical approval and should not have been reregistered or withdrawn.
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Shujun Li, Honorary Director of Nursing Department, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: 2024-IEC-0024-P-02
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Sleep; Newborn Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: All patients admitted to the neonatology department and neonatal intensive care unit were assessed for behavioral status using the Chinese version of the Neonatal Sleep-Wake Assessment Tool. Sleep cycles were also monitored using an electroencephalogram.

SUMMARY:
Sleep assessment of newborns in China is often neglected by medical staff, but sleep is related to the stability of vital signs and future neurobehavioral development. In order to understand the sleep quality of Chinese newborns and to protect their sleep during work, the neonatal sleep-wake assessment tool was translated into Chinese, revised, and tested for reliability and validity, in order to provide a reference for clinical staff to choose the timing of care.

ELIGIBILITY:
Inclusion Criteria:

* The clinical definition of a newborn was met.

Exclusion Criteria:

* A state of persistent convulsions

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates admitted to the department of Neonatology and neonatal intensive care unit who met the definition of newborn.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal sleep-wake state scores（composite outcome measure） | Results observed within 2 minutes.
  Behavioral state 4 items each scored and total score.The Chinese version of the Neonatal Sleep-Wake Assessment Tool included 4 items: eyes, breathing, facial expression, and movement. Each item was scored from 0 to 2 points, and the total score was from 0 to 8 points.Less than 3 points was defined as quiet sleep, 3-6 points as active sleep, and more than 6 points as awake sleep.

SECONDARY OUTCOMES:
Sleep state as shown by Amplitude-integrated EEG | Measurements were performed simultaneously with the Chinese version of the Neonatal Sleep-Wake Assessment Tool for 2minutes.
  The sleep-wake state of the newborn was obtained by aEEG analysis.The spectrum band of aEEG can be analyzed that the newborn is in a quiet sleep state, an active sleep state and an awake state. Generally, the narrow band refers to the awakening period and AS period, and the broad band refers to the QS period.

CONTACTS AND LOCATIONS:
Locations (1):
- CHZhejiang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided